CLINICAL TRIAL: NCT00234507
Title: Phase II, Multi-centre, Randomised, Double-blind, Parallel Group, Placebo-controlled Study to Assess the Efficacy and Safety of a Single Administration, by Subcutaneous Injection, of Three Doses of Dysport (40 Units/Eye, 80 Units/Eye, and 120 Units/Eye) for the Treatment of Benign Essential Blepharospasm
Brief Title: Study of a Single Administration of 3 Doses of Dysport® for the Treatment of Benign Essential Blepharospasm
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Y-47-52120-706
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Blepharospasm
MeSH Terms: conditions — Blepharospasm | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

INTERVENTIONS:
Biological: Botulinum toxin type A
  Other Names: AbobotulinumtoxinA (Dysport®)

SUMMARY:
The purpose of this study is to compare the effectiveness of 3 doses of Dysport® with placebo by assessing functional disability in blepharospasm.

ELIGIBILITY:
Inclusion Criteria:

* patients with a confirmed diagnosis of bilateral benign essential blepharospasm, and having symptoms of such for at least 6 months prior to the baseline visit
* naïve patients to botulinum toxin type A treatment, or patients who had received a single treatment of botulinum toxin type A, or those who had demonstrated a satisfactory response, in the investigator's opinion, to the last 2 injections of botulinum toxin type A with a minimum of 12 weeks since the last injection and where a further injection at full dosage was now indicated
* patients with a minimum score of 8 on the BDS

Exclusion Criteria:

* patients with either neuroleptic-induced blepharospasm, isolated levator dysfunction or apraxia
* previous surgical, chemical and thermal myectomy or neurectomy
* any condition where intramuscular injection is contraindicated
* ophthalmolgical infection
* myasthenia gravis or other disorders of the neuromuscular junction
* prescription of antispastic, muscle relaxants or medications affecting neuromuscular junction transmission, or medication where the dose or choice of medication has not been constant for the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2003-01; Primary Completion 2004-05-25 (Actual); Study Completion 2004-05-25 (Actual)

PRIMARY OUTCOMES:
The functional disability as measured by the percentage of normal activity (PNA) derived from the Blepharospasm Disability Scale (BDS) at 4 weeks post-treatment.

SECONDARY OUTCOMES:
Frequency of involuntary movements (FIM) and severity of oculo-facial spasm (measured by the Severity Rating Scale [SRS]) at 4 weeks post-treatment.
PNA, FIM and SRS at 8, 12 and 16 weeks post-treatment.
Severity of global impairment due to blepharospasm as measured by the Visual Analogue Scale (VAS) at 4, 8, 12 and 16 weeks post-treatment.
Change from baseline in BDS, FIM, severity of oculo-facial spasm and in severity of global impairment due to blepharospasm (measured by VAS) at 4, 8, 12 and 16 weeks post treatment.
Percentage of patients withdrawn from the study due to lack of efficacy at each assessment point.
Patient assessment of benefit and need for re-treatment, evaluated at the end of the study.
Investigator assessment of benefit and need for re-treatment, evaluated at the end of the study.
To compare the safety of each of the 3 doses of Dysport with placebo in terms of adverse event incidence, vital signs and physical examinations.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Study Director, Study Director — Ipsen
Locations (14):
- United States (14):
  - Banner Health Research Institute, Phoenix, Arizona
  - Neurological Institute, Phoenix, Arizona
  - The Parkinson's and Movement Disorder Institute, Fountain Valley, California
  - UCLA/Jules Stein Eye Institute, Los Angeles, California
  - McKnight Brain Institute, Gainesville, Florida
  - Plastic Eye Surgery Association, Pensacola, Florida
  - Rush Presbyterian/St Luke's Medical Center, Chicago, Illinois
  - Kellogg Eye Center, Ann Arbor, Michigan
  - Columbia-Presbyterian Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ophthlamic Surgeons and Consultants of Ohio, Inc, Columbus, Ohio
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Parkinson's Disease Center and Movement Disorders Clinic, Houston, Texas
  - Center for Facial Appearances, Salt Lake City, Utah